CLINICAL TRIAL: NCT01583478
Title: An Open-Label Pilot Study to Compare the Efficacy of Escalating Doses of IncobotulinumtoxinA (Xeomin®) in the Treatment of Glabellar Rhytids
Brief Title: Comparison of Escalating Doses of IncobotulinumtoxinA (Xeomin®) in the Treatment of Glabellar Rhytids
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Maas Clinic (Other)
Collaborators: Merz North America, Inc. (Industry)
Responsible Party: Principal Investigator, Corey S. Maas, M.D., Director, The Maas Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITGR-2012
Record Dates: First submitted 2012-03-20; First posted 2012-04-24 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Skin Aging; Elastosis Senilis
Keywords: incobotulinumtoxinA; wrinkles; glabellar; rhytids; frown; lines
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- incobotulinumtoxinA 20 units (Active Comparator): Three patients will be randomly assigned to receive 20 units total of incobotulinumtoxinA to the glabellar region.
  Interventions: Biological: incobotulinumtoxinA
- incobotulinumtoxinA 40 units (Active Comparator): Three patients will be randomly assigned to receive 40 units total of incobotulinumtoxinA to the glabellar region.
  Interventions: Biological: incobotulinumtoxinA
- incobotulinumtoxinA 60 units (Active Comparator): Three patients will be randomly assigned to receive 60 units total of incobotulinumtoxinA to the glabellar region.
  Interventions: Biological: incobotulinumtoxinA
- incobotulinumtoxinA 80 units (Active Comparator): Three patients will be randomly assigned to receive 80 units total of incobotulinumtoxinA to the glabellar region.
  Interventions: Biological: incobotulinumtoxinA
- incobotulinumtoxinA 100 units (Active Comparator): Three patients will be randomly assigned to receive 100 units total of incobotulinumtoxinA to the glabellar region.
  Interventions: Biological: incobotulinumtoxinA

INTERVENTIONS:
Biological: incobotulinumtoxinA — Eligible patients will receive Xeomin® doses of 20-, 40-, 60-, 80- or 100-units divided among 5 injection points (0.25 mL total) in the glabellar region on Day 0 of the study.
  Other Names: Xeomin®

SUMMARY:
The objective of the study is to compare the efficacy and duration of escalating doses of IncobotulinumtoxinA (Xeomin®) in the treatment of glabellar rhytids (frown lines between the eyes). Fifteen subjects will be enrolled in the study; specifically 60 male or female patients 18 years of age or older with moderate to severe glabellar rhytids at maximum contracture. Each patient will be randomized to receive one of 5 doses of Xeomin®, in a one-time dose to the treatment area.

The efficacy endpoints will be determined by investigator and subject live assessment of the glabellar rhytids at rest and maximum contraction at each visit (every other day for 6 days post-injection, every month for 9 months following) using a validated 4 point photographic scale (minimal wrinkles [0], mild wrinkles [1], moderate wrinkles [2], or severe wrinkles [3]) used in previous studies. A written description of each photograph will be included to help standardize the application of the Photographic Scale.

DETAILED DESCRIPTION:
Introduction Previously FDA-approved Botulinum type A toxins have been utilized in the upper face to treat glabellar rhytids for nearly two decades. Botox® Cosmetic (Allergan, Irvine, CA), is the first FDA-approved Botulinum toxin type A to be approved in the United States for the treatment of glabellar rhytids. Its efficacy and safety have been proven in multiple studies. Approximately two years ago, Dysport® (Medicis, Scottsdale, AZ) also received FDA approval for the treatment of dynamic glabellar rhytids. While both products have been on the market in Europe for over two decades, they have only been used in the United States for cosmetic applications for the past ten years. Xeomin® (Merz Pharmaceuticals, Frankfurt, Germany), at first, obtained FDA approval for the treatment of cervical dystonia and blepharospasm - two applications which the previous two botulinum type A toxins (onabotulinumtoxinA and abobotulinumtoxinA) had initially received prior to cosmetic approval. More recently, Xeomin® has been approved for cosmetic use. This study aims to assess the efficacy of varying doses of incobotulinumtoxinA in the treatment of glabellar rhytids.

Background Cosmetic procedures have been in increasing demand to reverse the appearance of advancing age, particularly procedures that improve the appearance of the aging face. Noninvasive procedures with little to no downtime that offer significant improvement to the aging appearance of the skin and underlying musculature are often preferred procedures to surgical options. Although no procedure is entirely risk free, continuing research is required to provide a safe and efficacious approach to aesthetic procedures for treating the aging face.

Although there are five factors that contribute to the appearance of the aging face,1 there are two anatomical units that most influence the appearance of facial rhytids: the skin and its underlying musculature. Many therapies have evolved to treat rhytids including resurfacing, topical preparations, soft tissue injectable fillers, and lastly, botulinum toxin.

Relaxation of facial musculature is routinely accomplished for cosmetic use by the use of Clostridium botulinum type A (BoNT-A). Clostridium botulinum type A toxin reduces the recruitment of specific muscle groups. Many studies have been published in peer-reviewed medical journals regarding the cosmetic use of this biologic.2-11 Clostridium botulinum in the form of Botox® Cosmetic (onabotulinumtoxinA) is FDA-approved for cosmetic use in the treatment of rhytids in the glabellar region. Dysport® (abobotulinumtoxinA) has been used similarly to treat the glabellar region received FDA approval in 2009. Xeomin® (incobotulinumtoxinA) received FDA approval in October 2010 for the treatment of cervical dystonia and blepharospasm, and has been used globally since 2005. Several studies have noted its efficacy in these clinical applications.12-16 More recently, Xeomin® (incobotulinumtoxinA) obtained FDA approval in July 2011 for cosmetic use. Its maker employs a manufacturing process which has isolated the active protein and eliminated accessory proteins present in other formulations.

Many studies have demonstrated the effect of botulinum toxin on facial rhytids produced by underlying coordinated muscle groups. Those of the glabellar area, upper forehead, lower forehead, periocular and perinasal area are particularly well-documented. Previous reports of Dysport® and Botox® Cosmetic medications show effective relaxation of glabellar rhytids after injection.12-17

Xeomin® is generally well-tolerated, although side effects may occur, such as temporary paralysis of adjacent muscle groups close to those injected, which may be due to local spread of toxin from the injection site and /or misplaced injections. Most side effects are mild or moderate severity, and of limited duration.

The most common adverse event (AE) seen following the use of Dysport®, Botox® Cosmetic or Xeomin® for the treatment of blepharospasm is ptosis. Some patients have reported diplopia or symptoms resulting from the spread of effect to mid-facial muscles. Other AEs reported were injection site reaction, skin rashes, influenza-like symptoms, dry eyes, tearing, bruising, and eyelid swelling. Reversible ophthalmoplegia has been reported after excessive dosing.

Studies have shown safety of high doses of botulinum toxin type A for the treatment of spasticity and hyperhydrosis in both children and adults with doses ranging from 400 to upwards of 1200 units in a single-dose injection.18,19

No clinical studies have been conducted in North America to determine the optimal dosing of Xeomin® for cosmetic use in the glabellar area. Though the manufacturers of Xeomin® purported a 1:1 dosage ratio with Botox® Cosmetic, this conversion has not been demonstrated or proven in facial cosmetic applications. This study intends to compare varying doses of incobotulinumtoxinA in the treatment of glabellar rhytids to assess which dosage is the most optimal in terms of efficacy and duration of action.

Investigational Agents Xeomin® is supplied as a 100 unit vial of Clostridium botulinum type A exotoxin, sterilely prepared and vacuum-dried without preservatives.

Dose Rationale and Risk/Benefits:

Administration Eligible patients will receive Xeomin® doses of escalating-units divided among 5 injection points (0.25 mL total) in the glabellar region on Day 0 of the study, as described in the instructions section.

For Study Purposes:

For study purposes, only one injection session will be performed at Day 0 of the study. Subsequent follow-up visits will only monitor the effects of the single injection session at time 0.

Packaging, Labeling, and Storage Commercially-available active drug (Xeomin®) vials, bearing a unique lot number, will be obtained from Merz Pharmaceuticals.

Study medications may be maintained during transit and storage within a temperature range of 20o to 25o C, refrigerated within a temperature range of 2o to 8o C or frozen within a temperature range of -20o to -10o C.

Drug accountability The investigator will administer study medication only to patients included in this study and following the procedures set out in this study protocol. Each dispensing will be documented in the CRFs and the study medication dispensing log.

Concomitant Medications and Treatments Any medication the patient takes other than the study medication specified in the protocol is considered a concomitant medication. This applies to prescription and over-the-counter (OTC) drugs, and to herbal supplements, whether taken systemically or applied topically. In addition, any treatment the patient receives other than the study medication is considered a concomitant treatment. This applies to cosmetic treatments of the face and neck area. All concomitant medications and concomitant treatments must be recorded in the CRFs.

Prohibited medication classes and treatments are described under "Exclusion Criteria". In the event that a prohibited treatment (e.g. microdermabrasion, Intense Pulse Light, light-emitting diodes, or radio-frequency) is received, it must be documented on the CRFs.

Study Objectives

Primary Objective:

To compare the efficacy of escalating doses of Xeomin® in the treatment of glabellar rhytids.

Secondary Objective:

To assess the duration of action of escalating doses of Xeomin® in the treatment of glabellar rhytids.

Secondary Objective:

To determine the safety and presence of any adverse effects of Xeomin® in the treatment of glabellar rhytids.

Study Design General Design

* Phase IV, single-center, prospective, open-label study.
* 60 subjects with moderate to severe glabellar rhytids.
* 12 month duration
* 16 Visits: Visit 0 Screening/Baseline(treatment), Visit 1 follow-up (day 1), Visit 2 follow-up (day 4), Visit 3 follow-up (day 7), Visit 4 (day 30), Visit 5 (day 60), Visit 6 (day 90), Visit 7 (day 120), Visit 8 (day 150), Visit 9 (day 180), Visit 10 (day 210), Visit 11 (day 240), Visit 12 (day 270), Visit 13 (day 300), Visit 14 (day 330), Visit 15 (day 360). If patients are assessed and have returned to baseline at any visit prior to Visit 15, then they will be seen at their next two sequential follow-up visits to allow for any possible variations in assessment or adverse events.

Primary Study Endpoints

Efficacy and duration endpoints will be determined by:

* The investigator's live assessment of glabellar rhytids at maximum contraction and at rest.

Secondary adverse event endpoints will be determined by:

* The patient's assessment of any symptoms experienced between follow-up visits as recorded on the CRF.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients who meet all of the following criteria are eligible for this study:

* Eighteen years of age or older.
* Moderate to severe vertical glabellar lines at maximum frown (score of [2] or [3] by physician assessment)
* Negative pregnancy test for females of childbearing potential.
* Time and ability to complete the study and comply with instructions.
* Understanding of the study and contents of the informed consent.

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for this study:

* Previous treatment to the glabellar area with Dysport® or Botox® Cosmetic or other botulinum toxin within 90 days of entry into the study. Botulinum toxin treatment of areas other than the glabellar area at any time during the study.
* Patients with an ongoing treatment-related AE from any Dysport® or Botox® Cosmetic or botulinum toxin study.
* Inability to substantially lessen glabellar lines by physically spreading them apart.
* Soft tissue augmentation of the glabellar area (e.g. collagen-type implants, or hyaluronic acid fillers) at any time during the current study.
* Permanent or semi-permanent dermal fillers in the glabellar area at any time.
* Ablative skin resurfacing on the glabellar area at any time preceding the study or planning to during the current study.
* Upper eyelid blepharoplasty or brow-lift at any time preceding the study or planning to during the current study.
* Non-ablative treatments in the glabellar area for skin dyschromias (e.g. Intense Pulsed Light, light-emitting diodes) at any time during the current study.
* Non-ablative dermal treatment in the glabellar area for skin tightening (e.g. radiofrequency treatments at any time preceding the current study or plan to have this done during the current study)
* Retinoid, microdermabrasion, or prescription-level glycolic acid treatments to the glabellar area within 2 weeks prior to study participation or during the current study.
* Concurrent therapy that, in the investigator's opinion, would interfere with evaluation of the efficacy or safety of the medication.
* Active infection of the glabellar area (e.g. acute acne lesions or ulcers).
* Pregnant women, nursing mothers, or women who are planning pregnancy during the study, or think they may be pregnant at the start of the study. Throughout the course of the study, women of childbearing potential must use reliable forms of contraception (e.g. abstinence, oral contraceptives for more than 12 consecutive weeks prior to enrollment, or spermicide and condoms).
* Current history of chronic drug or alcohol abuse.
* Enrollment in any active study involving the use of investigational devices or drugs.
* Current facial palsy.
* Marked facial asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin.
* Neuromuscular junctional disorders (myasthenia gravis).
* Known allergy or hypersensitivity to any botulinum toxin or any component of Dysport® or Botox® Cosmetic.
* Clinically diagnosed anxiety disorder, or any other significant psychiatric disorder (e.g. depression) that, in the opinion of the investigator, might interfere with the patient's participation in the study.
* Concurrent use of medications that affect neuromuscular transmission, such as curare-like depolarizing agents, lincosamides, polymyxins, anticholinesterases affecting the striated muscle, and aminoglycoside antibiotics.
* Presence of any condition (e.g. neuromuscular disorder or other disorder that could interfere with neuromuscular function) or circumstance that, in the judgment of the investigator, might increase the risk to the patient or decrease the chance of obtaining satisfactory data to achieve the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of escalating doses of Xeomin® in the treatment of glabellar rhytids | 12 months
  Investigator and subject assessed grading

SECONDARY OUTCOMES:
Duration of action of escalating doses of Xeomin® in the treatment of glabellar rhytids | 12 months
  Investigator and subject assessed grading
Safety and presence of any adverse effects of Xeomin® in the treatment of glabellar rhytids | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Corey S Maas, MD, Principal Investigator — The Maas Clinic
Locations (1):
- The Maas Clinic, San Francisco, California, United States